CLINICAL TRIAL: NCT02561078
Title: Safety and Efficacy of Human Regular U-500 Insulin Administered by Continuous Subcutaneous Insulin Infusion Versus Multiple Daily Injections in Subjects With Type 2 Diabetes Mellitus: A Randomized, Open-Label, Parallel Clinical Trial
Brief Title: An Administration Method Study of Human Regular U-500 Insulin (LY041001) in Participants With Type 2 Diabetes Mellitus
Acronym: VIVID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Insulet Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14902; B5K-MC-IBHD (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-09-23; First posted 2015-09-25 (Estimated); Results first posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: insulin pumps; concentrated insulin; OmniPod
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Human regular U-500 insulin administered by CSII (Experimental): Human regular U-500 insulin administered by CSII and titrated based on blood glucose readings for 26 weeks with a 2-week MDI lead-in.
  Interventions: Drug: Human regular U-500 insulin (CSII)
- Human regular U-500 insulin administered by MDI (Active Comparator): Human regular U-500 insulin administered subcutaneously (SC) by MDI three times a day and titrated based on blood glucose readings for 26 weeks.
  Interventions: Drug: Human regular U-500 insulin (MDI)

INTERVENTIONS:
Drug: Human regular U-500 insulin (CSII) — Administered SC
  Other Names: LY041001
  Arms: Human regular U-500 insulin administered by CSII
Drug: Human regular U-500 insulin (MDI) — Administered SC
  Other Names: LY041001
  Arms: Human regular U-500 insulin administered by MDI

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of the study drug known as human regular U-500 insulin (U-500R) administered by continuous subcutaneous insulin infusion (CSII) versus multiple daily injections (MDI) in participants with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes mellitus (T2DM).
* Current TDD >200 but ≤600 units of non U-500R insulin (MDI or CSII) and/or U-500R by MDI with syringe and vial for ≥3 months at entry.

  * If TDD of U-500R and other insulins are combined, then insulin other than U-500R not to exceed 25% of TDD.
* HbA1c ≥7.5% and ≤12.0%.
* Body mass index ≥25 but ≤50 kilograms per meter squared.
* Have a history of stable body weight.
* Concomitant antihyperglycemic agent (AHA) therapy may include metformin (MET), dipeptidyl peptidase-4 inhibitors and/or pioglitazone.

  * Approximately 64 to 96 subjects using glucagon-like peptide-1 (GLP-1) receptor agonists or sodium-glucose cotransporter 2 (SGLT2) inhibitors will be enrolled in Study Group B.

Exclusion Criteria:

* Diagnosed with type 1 diabetes mellitus (T1DM) or other types of diabetes apart from T2DM.
* Have obvious clinical or radiographic signs or symptoms of liver disease (except nonalcoholic fatty liver disease), cirrhosis, acute or chronic hepatitis, or alanine aminotransferase (ALT/SGPT) and/or aspartate aminotransferase (AST/SGOT) levels ≥2.5X upper limit of normal (ULN), alkaline phosphatase ≥2X ULN or total bilirubin ≥2X ULN.
* Have chronic kidney disease Stage 4 and higher or history of renal transplantation.
* Have history of more than 1 episode of severe hypoglycemia within the 6 months prior to screening.
* Have received U-500R insulin by CSII in the 3 months prior to screening.
* Have had a blood transfusion or severe blood loss within 3 months prior to screening or have known hemoglobinopathy, hemolytic anemia, or sickle cell anemia.
* Are taking chronic (lasting longer than 14 consecutive days) systemic glucocorticoid therapy.
* Have an irregular sleep/wake cycle.
* Have used any weight loss drugs in the 3 months prior to screening.
* Have a history of bariatric surgery including Roux-en-Y gastric bypass surgery, gastric banding, and/or gastric sleeve.
* Have a history of an active or untreated malignancy, or in remission from a clinically significant malignancy during the last 5 years before screening.
* Significant hearing loss and/or vision impairment deemed by the investigator to interfere with the safe use of OmniPod U-500 system.
* Have cardiac disease with functional status that is New York Heart Association (NYHA) Class III or IV per New York Heart Association Cardiac Disease Functional Classification or have congestive heart failure requiring pharmacologic treatment.
* Are women breastfeeding or pregnant, or intend to become pregnant during the course of the study; are men who intend to impregnate their partners; or are sexually active of procreation potential not actively practicing birth control by a method determined by the investigator to be medically acceptable. Are investigator site personnel directly affiliated with this study and/or their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2017-05-09 (Actual); Study Completion 2017-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (56):
- United States (51):
  - Internal Medicine Center LLC, Mobile, Alabama
  - John Muir Physician Network Clinical Research Center, Concord, California
  - Valley Endocrine, Fresno, Fresno, California
  - Scripps Whittier Diabetes Institute, La Jolla, California
  - Diabetes and Endocrine Associates, La Mesa, California
  - First Valley Medical Group, Lancaster, California
  - Pacific Research Partners, LLC, Oakland, California
  - Inland Empire Liver Foundation, Rialto, California
  - NorCal Endocrinology and Internal Medicine - Roseville, Roseville, California
  - NorCal Endocrinology and Internal Medicine - Roseville, San Ramon, California
  - Olive View Medical Center, Sylmar, California
  - ALL Medical Research, LLC, Cooper City, Florida
  - East Coast Institute For Research, LLC, Jacksonville, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Metabolic Research Institute Inc., West Palm Beach, Florida
  - East Coast Institute For Research, LLC, Macon, Georgia
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - John H. Stroger Hospital of Cook County, Chicago, Illinois
  - Midwest CRC, Crystal Lake, Illinois
  - HSHS Medical Group Diabetes Research, Springfield, Illinois
  - Iderc, P.L.C., Des Moines, Iowa
  - Cotton O'Neil Diabetes and Endocrinology Center, Topeka, Kansas
  - Kentucky Diabetes Endocrinology Center, Lexington, Kentucky
  - The Arthritis & Diabetes Clinic Inc., Monroe, Louisiana
  - Grunberger Diabetes Institute, Bloomfield Hills, Michigan
  - Adult Endocrinology Consultants, P.C., Livonia, Michigan
  - JCMG Clinical Research, Jefferson City, Missouri
  - Billings Clinic Research Center, Billings, Montana
  - Diabetes and Endocrinology Associates, Omaha, Nebraska
  - Palm Research Center, Las Vegas, Nevada
  - Southern New Hampshire Diabetes and Endocrinology, Nashua, New Hampshire
  - North Shore Diabetes and Endocrine Assoc, New Hyde Park, New York
  - Mountain Diabetes and Endocrine Center, Asheville, North Carolina
  - Physicians East, Greenville, North Carolina
  - PMG Research of Rocky Mount, LLC, Rocky Mount, North Carolina
  - University of Oklahoma Health Sciences Center-Tulsa, Oklahoma City, Oklahoma
  - Portland Diabetes & Endocrine Center, Portland, Oregon
  - Endocrine Metabolic Associates, P.C., Philadelphia, Pennsylvania
  - Partners in Nephrology & Endocrinology, Pittsburgh, Pennsylvania
  - Sudhir Bansal M.D. Inc., Warwick, Rhode Island
  - AM Diabetes and Endocrinology Center, Bartlett, Tennessee
  - University Diabetes and Endocrine Consultants, Chattanooga, Tennessee
  - Vanderbilt Univeristy School of Medicine, Nashville, Tennessee
  - Texas Diabetes and Endocrinology-Austin South, Austin, Texas
  - Dallas Diabetes Endocrine Center, Dallas, Texas
  - Texas Diabetes and Endocrinology, P.A., Round Rock, Texas
  - Advanced Research Institute, South Ogden, Utah
  - Dr. Larry Stonesifer, Federal Way, Washington
  - Rainier Clinical Research Center, Renton, Washington
  - Northside Internal Medicine, Spokane, Washington
  - Multicare Health System, Tacoma, Washington
- Puerto Rico (5):
  - Dr Altagracia Aurora Alcantara Gonzalez, Bayamón
  - Manati Center for Clinical Research Inc, Manatí
  - Endocrine Lipid Diabetes Research Institute, Ponce
  - American Telemedicine Center, San Juan
  - Martha Gomez Cuellar M.D., San Juan

REFERENCES:
- See also: Click here for more information about this study: An Administration Method Study of Human Regular U-500 Insulin (LY041001) in Participants With Type 2 Diabetes Mellitus — https://www.lillytrialguide.com/en-US/studies/adult-type-2-diabetes/IBHD#?postal=

RESULTS

PARTICIPANT FLOW:
Groups:
- Human Regular U-500 Insulin Administered by CSII: Human regular U-500 insulin administered by continuous subcutaneous insulin infusion (CSII) and titrated based on blood glucose readings for 26 weeks with a 2-week multiple daily injections (MDI) lead-in.
- Human Regular U-500 Insulin Administered by MDI: Human regular U-500 insulin administered subcutaneously (SC) by multiple daily injections (MDI) three times a day and titrated based on blood glucose readings for 26 weeks.
Period: Overall Study
Arm/Group | Human Regular U-500 Insulin Administered by CSII | Human Regular U-500 Insulin Administered by MDI
Started | 209 | 211
Received at Least 1 Dose of Study Drug | 208 | 210
Completed | 179 | 186
Not Completed | 30 | 25
Not completed — Adverse Event | 5 | 2
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 2 | 6
Not completed — Non-Compliance with Study Drug | 6 | 3
Not completed — Physician Decision | 2 | 3
Not completed — Withdrawal by Subject | 13 | 10

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Human Regular U-500 Insulin Administered by CSII | Human Regular U-500 Insulin Administered by MDI | Total
Number analyzed (Participants) | 209 | 211 | 420
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.58 (10.27) | 56.66 (10.12) | 57.12 (10.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 94 | 199
  Male | 104 | 117 | 221
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 49 | 88
  Not Hispanic or Latino | 170 | 162 | 332
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 2 | 7 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 19 | 14 | 33
  White | 160 | 160 | 320
  More than one race | 25 | 26 | 51
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 15 | 21 | 36
  United States | 194 | 190 | 384
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.
  Percentage of HbA1c | 8.75 (1.03) | 8.77 (1.08) | 8.76 (1.05)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.
  Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with baseline of response, glucagon-like peptide-1 (GLP-1) or sodium-glucose cotransporter 2 (SGLT2) use, U-500R at entry, treatment, time and treatment by time interaction.
Time Frame: Baseline, 26 Weeks
Population: All randomized participants who received at least 1 dose of study drug with baseline and post-baseline HbA1c measure.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Human Regular U-500 Insulin Administered by CSII | Human Regular U-500 Insulin Administered by MDI
Number analyzed (Participants) | 171 | 179
Percentage of HbA1c | -1.27 (0.072) | -0.85 (0.070)
Statistical Analysis 1: Comparison: Human Regular U-500 Insulin Administered by CSII vs Human Regular U-500 Insulin Administered by MDI; Test type: Non-Inferiority — The test for the primary objective of noninferiority was performed at the 0.05 significance level using the LS Mean estimate of the difference in change in HbA1c between the 2 treatments at Week 26. Noninferiority was established if the upper limit of a 2-sided 95% confidence interval (CI) for the difference (U 500R CSII minus U 500R MDI) was below the noninferiority margin (NIM) of 0.4%; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.42, 95% CI 2-sided [-0.62 to -0.22]

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Fasting plasma glucose (FPG) is a test to determine how much glucose (sugar) is in a plasma sample after an overnight fast. Least Squares (LS) means was determined by MMRM methodology with baseline of response, glucagon-like peptide-1 (GLP-1) or sodium-glucose cotransporter 2 (SGLT2) use, U-500R at entry, treatment, time and treatment by time interaction.
Time Frame: Baseline, 26 Weeks
Population: All randomized participants who received at least 1 dose of study drug with baseline and post-baseline fasting plasma glucose measure.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | Human Regular U-500 Insulin Administered by CSII | Human Regular U-500 Insulin Administered by MDI
Number analyzed (Participants) | 163 | 172
milligrams per deciliter (mg/dL) | -33.9 (5.03) | 1.7 (4.90)
Statistical Analysis 1: Comparison: Human Regular U-500 Insulin Administered by CSII vs Human Regular U-500 Insulin Administered by MDI; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -35.6, 95% CI 2-sided [-49.4 to -21.7]

3. Secondary Outcome: Percentage of Participants With HbA1c <7.0%
Description: Hemoglobin A1c (HbA1c) is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. Longitudinal logistic regression was used to model the likelihood of having hbA1c<7.0% at Week 26 with baseline of response, glucagon-like peptide-1 (GLP-1) or sodium-glucose cotransporter 2 (SGLT2) use, U-500R at entry, treatment, time and treatment by time interaction.
Time Frame: 26 Weeks
Population: All randomized participants who received at least 1 dose of study drug with baseline and post-baseline HbA1c measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Human Regular U-500 Insulin Administered by CSII | Human Regular U-500 Insulin Administered by MDI
Number analyzed (Participants) | 171 | 179
Percentage of participants | 28.65 | 18.44
Statistical Analysis 1: Comparison: Human Regular U-500 Insulin Administered by CSII vs Human Regular U-500 Insulin Administered by MDI; Test type: Superiority; p = 0.015, Regression, Logistic; Odds Ratio (OR) = 1.97, 95% CI 2-sided [1.14 to 3.39]

4. Secondary Outcome: Percentage of Participants With HbA1c <7.5%
Description: Hemoglobin A1c (HbA1c) is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. Longitudinal logistic regression was used to model the likelihood of having hbA1c<7.5% at Week 26 with baseline of response, glucagon-like peptide-1 (GLP-1) or sodium-glucose cotransporter 2 (SGLT2) use, U-500R at entry, treatment, time and treatment by time interaction.
Time Frame: 26 Weeks
Population: All randomized participants who received at least 1 dose of study drug with baseline and post-baseline HbA1c measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Human Regular U-500 Insulin Administered by CSII | Human Regular U-500 Insulin Administered by MDI
Number analyzed (Participants) | 171 | 179
Percentage of Participants | 52.63 | 38.55
Statistical Analysis 1: Comparison: Human Regular U-500 Insulin Administered by CSII vs Human Regular U-500 Insulin Administered by MDI; Test type: Superiority; p = 0.005, Regression, Logistic; Odds Ratio (OR) = 1.94, 95% CI 2-sided [1.23 to 3.07]

5. Secondary Outcome: Change From Baseline in 7-point Self-Monitored Blood Glucose (SMBG) Values
Description: Seven-point SMBG are completed at the following timepoints: Before Morning Meal, 2 Hours After Morning Meal, Before Mid-Day Meal, 2 Hours After Mid-Day Meal, Before Evening Meal, Bed Time and 03:00 AM hours. Least Squares (LS) means was determined by mixed model repeated measures (MMRM) methodology with baseline of response, GLP-1 or SGLT2 use, U-500R at entry, baseline HbA1C group, treatment, time and treatment by time interaction.
Time Frame: Baseline, 26 Weeks
Population: All randomized participants who received at least 1 dose of study drug with baseline and post-baseline SMBG measure.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Human Regular U-500 Insulin Administered by CSII | Human Regular U-500 Insulin Administered by MDI
Number analyzed (Participants) | 140 | 151
mg/dL
  Pre Morning Meal: number analyzed (Participants) | 139 | 150
  Pre Morning Meal | -34.3 (3.53) | -11.8 (3.41)
  2 Hours Post Morning Meal: number analyzed (Participants) | 129 | 136
  2 Hours Post Morning Meal | -25.0 (4.58) | -7.8 (4.50)
  Pre Mid-Day Meal: number analyzed (Participants) | 139 | 151
  Pre Mid-Day Meal | -19.8 (4.29) | -10.9 (4.15)
  2 Hours Post Mid-Day Meal: number analyzed (Participants) | 129 | 138
  2 Hours Post Mid-Day Meal | -8.3 (4.20) | -16.6 (4.08)
  Pre Evening Meal: number analyzed (Participants) | 140 | 149
  Pre Evening Meal | -15.1 (4.11) | -24.3 (3.99)
  2 HOURS POST EVENING MEAL: number analyzed (Participants) | 134 | 147
  2 HOURS POST EVENING MEAL | -14.6 (4.19) | -31.3 (4.02)
  OVERNIGHT (3:00 AM): number analyzed (Participants) | 121 | 127
  OVERNIGHT (3:00 AM) | -25.4 (3.71) | -26.0 (3.58)
Statistical Analysis 1: Comparison: Human Regular U-500 Insulin Administered by CSII vs Human Regular U-500 Insulin Administered by MDI; Pre Morning Meal; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -22.5, 95% CI 2-sided [-32.1 to -12.8]
Statistical Analysis 2: Comparison: Human Regular U-500 Insulin Administered by CSII vs Human Regular U-500 Insulin Administered by MDI; 2 Hours Post Morning Meal; Test type: Superiority; p = 0.008, Mixed Models Analysis; Mean Difference (Net) = -17.2, 95% CI 2-sided [-29.9 to -4.6]
Statistical Analysis 3: Comparison: Human Regular U-500 Insulin Administered by CSII vs Human Regular U-500 Insulin Administered by MDI; Pre Mid-Day Meal; Test type: Superiority; p = 0.138, Mixed Models Analysis; Mean Difference (Net) = -8.9, 95% CI 2-sided [-20.6 to 2.9]
Statistical Analysis 4: Comparison: Human Regular U-500 Insulin Administered by CSII vs Human Regular U-500 Insulin Administered by MDI; 2 Hours Post Mid-Day Meal; Test type: Superiority; p = 0.160, Mixed Models Analysis; Mean Difference (Net) = 8.3, 95% CI 2-sided [-3.3 to 19.8]
Statistical Analysis 5: Comparison: Human Regular U-500 Insulin Administered by CSII vs Human Regular U-500 Insulin Administered by MDI; Pre Evening Meal; Test type: Superiority; p = 0.113, Mixed Models Analysis; Mean Difference (Net) = 9.1, 95% CI 2-sided [-2.2 to 20.4]
Statistical Analysis 6: Comparison: Human Regular U-500 Insulin Administered by CSII vs Human Regular U-500 Insulin Administered by MDI; 2 Hours Post Evening Meal; Test type: Superiority; p = 0.004, Mixed Models Analysis; Mean Difference (Net) = 16.7, 95% CI 2-sided [5.3 to 28.2]
Statistical Analysis 7: Comparison: Human Regular U-500 Insulin Administered by CSII vs Human Regular U-500 Insulin Administered by MDI; Overnight (3:00 AM); Test type: Superiority; p = 0.905, Mixed Models Analysis; Mean Difference (Net) = 0.6, 95% CI 2-sided [-9.5 to 10.8]

6. Secondary Outcome: Change From Baseline in Total Daily Dose (TDD)
Description: Baseline TDD was defined as the last prestudy insulin TDD prior to randomization to receiving the first dose of U-500 insulin post randomization. Least Squares (LS) means was determined by mixed model repeated measures (MMRM) methodology with baseline of response, GLP-1 or SGLT2 use, U-500R at entry, baseline HbA1C group, treatment, time and treatment by time interaction.
Time Frame: Baseline, 26 Weeks
Population: All randomized participants who received at least 1 dose of study drug with baseline and post-baseline TDD measure.
Measure: Least Squares Mean (Standard Error); unit: units/day
Arm/Group | Human Regular U-500 Insulin Administered by CSII | Human Regular U-500 Insulin Administered by MDI
Number analyzed (Participants) | 172 | 180
units/day | 2.8 (9.33) | 51.3 (9.14)
Statistical Analysis 1: Comparison: Human Regular U-500 Insulin Administered by CSII vs Human Regular U-500 Insulin Administered by MDI; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -48.4, 95% CI 2-sided [-74.1 to -22.8]

7. Secondary Outcome: Percentage of Participants With Hypoglycemic Episodes (Documented Hypoglycemia With Blood Glucose <= 70 mg/dL)
Description: The percentage of participants with hypoglycemic episodes (documented hypoglycemia) was calculated by dividing the number of participants with at least 1 hypoglycemic episode (documented hypoglycemia) over the 26-week treatment period by the total number of participants analyzed, multiplied by 100%. Logistic regression was used to estimate the odds ratio between the two treatments of at least 1 hypoglycemic episode (documented hypoglycemia) over 26 week treatment period adjusted for baseline documented hypoglycemia rate, GLP-1 or SGLT2 use, U-500R at entry, baseline HbA1C group, treatment, time and treatment by time interaction.
Time Frame: 26 Weeks
Population: All randomized participants who received at least 1 dose of study drug with baseline and post-baseline documented hypoglycemia.
Measure: Number; unit: Percentage of Participants
Arm/Group | Human Regular U-500 Insulin Administered by CSII | Human Regular U-500 Insulin Administered by MDI
Number analyzed (Participants) | 209 | 210
Percentage of Participants | 95.69 | 95.71
Statistical Analysis 1: Comparison: Human Regular U-500 Insulin Administered by CSII vs Human Regular U-500 Insulin Administered by MDI; Test type: Superiority; p = 0.919, Regression, Logistic; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.39 to 2.86]

8. Secondary Outcome: Rate of Hypoglycemic Episodes (Documented Hypoglycemia With Blood Glucose <= 70 mg/dL)
Description: Documented Hypoglycemic episodes with blood glucose<=70mg/dL was used in this outcome measure. Hypoglycemia rate (documented hypoglycemia) per 30 days was summarized at each visit by treatment group. The rate of hypoglycemia (documented hypoglycemia) was analyzed using a generalized estimation equations model with a negative binomial distribution and a Log link. LS mean was determined by MMRM methodology with baseline documented hypoglycemia rate, GLP-1 or SGLT2 use, U-500R at entry, baseline HbA1C group, with log of exposure in days divided by 30 as the offset, treatment, visit, and visit by treatment interaction.
Time Frame: Baseline to 26 Weeks
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Episodes/participant/30 days
Arm/Group | Human Regular U-500 Insulin Administered by CSII | Human Regular U-500 Insulin Administered by MDI
Number analyzed (Participants) | 209 | 210
Episodes/participant/30 days | 5.16 (0.380) | 4.27 (0.308)
Statistical Analysis 1: Comparison: Human Regular U-500 Insulin Administered by CSII vs Human Regular U-500 Insulin Administered by MDI; Test type: Superiority; p = 0.025, Negative binomial regression; Relative Rate = 1.21, 95% CI 2-sided [1.02 to 1.42]

9. Secondary Outcome: Change From Baseline in Body Weight
Description: Least Squares (LS) means was determined by mixed model repeated measures (MMRM) methodology with baseline of response, GLP-1 or SGLT2 use, U-500R at entry, baseline HbA1C group, treatment, treatment by time interaction.
Time Frame: Baseline, 26 Weeks
Population: All randomized participants who received at least 1 dose of study drug with baseline and post-baseline body weight.
Measure: Least Squares Mean (Standard Error); unit: Kilograms (kg)
Arm/Group | Human Regular U-500 Insulin Administered by CSII | Human Regular U-500 Insulin Administered by MDI
Number analyzed (Participants) | 171 | 181
Kilograms (kg) | 4.2 (0.35) | 3.4 (0.34)
Statistical Analysis 1: Comparison: Human Regular U-500 Insulin Administered by CSII vs Human Regular U-500 Insulin Administered by MDI; Test type: Superiority; p = 0.100, Mixed Models Analysis; Mean Difference (Net) = 0.8, 95% CI 2-sided [-0.2 to 1.8]

ADVERSE EVENTS:
Time Frame: Up to 26 weeks
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Human Regular U-500 Insulin Administered by CSII | Human Regular U-500 Insulin Administered by MDI
All-Cause Mortality (participants affected / at risk) | 2/209 | 1/211
Serious Adverse Events (participants affected / at risk) | 34/209 | 23/211
Other Adverse Events (participants affected / at risk) | 85/209 | 84/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human Regular U-500 Insulin Administered by CSII (N=209) | Human Regular U-500 Insulin Administered by MDI (N=211)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Cor pulmonale (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 10 (12) | 5 (5)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Moyamoya disease (Nervous system disorders) | 1 (1) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 3 (3)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human Regular U-500 Insulin Administered by CSII (N=209) | Human Regular U-500 Insulin Administered by MDI (N=211)
Diarrhoea (Gastrointestinal disorders) | 14 (18) | 17 (22)
Nausea (Gastrointestinal disorders) | 9 (9) | 17 (20)
Sinusitis (Infections and infestations) | 10 (10) | 13 (15)
Upper respiratory tract infection (Infections and infestations) | 17 (17) | 18 (19)
Urinary tract infection (Infections and infestations) | 3 (4) | 11 (11)
Viral upper respiratory tract infection (Infections and infestations) | 11 (12) | 18 (21)
Weight increased (Investigations) | 14 (14) | 13 (13)
Hyperglycaemia (Metabolism and nutrition disorders) | 11 (17) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 13 (16)
Headache (Nervous system disorders) | 9 (11) | 14 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 12 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (3):
  • Study Protocol: Study Protocol (2015-06-11): https://cdn.clinicaltrials.gov/large-docs/78/NCT02561078/Prot_003.pdf
  • Statistical Analysis Plan (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/78/NCT02561078/SAP_004.pdf
  • Study Protocol: Study Protocol (a) (2016-12-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT02561078/Prot_005.pdf